CLINICAL TRIAL: NCT04780594
Title: Impact of the SARS-CoV-2 (COVID-19) Pandemic on the Morbidity and Mortality of Patients Undergoing Surgery at Bellvitge University Hospital
Brief Title: Impact of the COVID-19 Pandemic on the Surgical Activity of Bellvitge University Hospital
Status: Completed | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Marta Caballero Milan, Medical Staff in Anaesthesiology and Reanimation, Hospital Universitari de Bellvitge
Other Study IDs: COVID19 surgical impact
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Surgery--Complications; Nosocomial Infection
Keywords: COVID19; Hospital stay; mortality; surgery complications; scheduled surgery; emergency surgery
MeSH Terms: conditions — COVID-19; Cross Infection

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-pandemic COVID-19 group (PreCOVID): All patients who underwent surgery from 13th January until 29th February 2020, which are considered free of COVID-19 patients, therefore pre-pandemic period.
  Interventions: Procedure: The study evaluates all surgical patients operated, both elective scheduled and emergent cases
- Pandemic COVID-19 group (COVID): All patients who underwent surgery from 11th March 2020 until 15th May 2020, which were done during the first wave of the pandemic crisis.
  Interventions: Procedure: The study evaluates all surgical patients operated, both elective scheduled and emergent cases

INTERVENTIONS:
Procedure: The study evaluates all surgical patients operated, both elective scheduled and emergent cases — Administrative database was automatically collected. That included demographic, clinical antecedents, surgical team and surgical procedure, primary and secondary diagnoses and principal and secondary surgical procedures. A case-mix grouping system administrative automatic recorded based on the ICD-10-AM International Classification of Diseases. According to the Diagnoses-related Groups (DRG's). the Severity of Illness Index assigns to each patient an overall severity score (from 1 to 4) and mortality risk score (from 1 to 4)

SUMMARY:
COVID-19 has been a challenge for hospitals; there was an obvious need to reconvert many spaces in specific areas to attend this pathology, without forgetting the attention to other pathologies and surgery. The objective of the investigators is to evaluate the impact of this pandemic in the patients who underwent surgery in Bellvitge University Hospital, analyzing 2 periods of time: the months before the COVID-19 peak and the COVID-19 peak months.

DETAILED DESCRIPTION:
A total of 2.530 procedures have been evaluated in this retrospective observational study. Two groups have been generated (pre-pandemic period and pandemic period), classified into scheduled and emergency surgery. The investigators determined age, type of surgery and specialty, hospital stay, destination at discharge including mortality and severity according to Diagnostic Related to Group (DRG) scale. The investigators have also determined the number of confirmed COVID-19 infections in patients who underwent surgery during these 2 periods and evaluated if the infection was due to a nosocomial infection (confirmation of the COVID-19 during the hospitalization period). Comparisons were made between subgroups: scheduled surgery performed during the 2 periods and emergency surgery performed during the 2 periods.

ELIGIBILITY:
Inclusion Criteria:

* All surgical patients operated, both elective scheduled and emergent cases

Exclusion Criteria:

* Minor-intermediate surgery that involves discharge from the hospital on the same day of the surgery from the Pre-pandemic period.
* Procedures related to medical treatment or complications of COVID-19 patients, such as chest tubes, extracorporeal oxygenation or tracheostomy.
* Those scheduled elective surgery patients in the Covid period that resulted RT-PCR positive, surgery was posponed, were not considered eligible for the analysis.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The requirement to include patients was that they required surgery, either urgent or scheduled, during the periods described (PreCOVID and COVID). As there is no paediatric service in the hospital, the minimum age of the sample is 18 years old but there is no maximum age for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 2530 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Register the post-surgical complications | PreCOVID group from 13th January 2020 to 29th February 2020 and COVID group from 11th March 2020 to 15th May 2020.
  Register and Compare the Rate of Surgical Reintervention between both periods.

SECONDARY OUTCOMES:
Register the rate of surgical reintervention | PreCOVID group from 13th January 2020 to 29th February 2020 and COVID group from 11th March 2020 to 15th May 2020.
  Register and compare the Rate of reintervention between both periods.
Register the ICU admission | PreCOVID group from 13th January 2020 to 29th February 2020 and COVID group from 11th March 2020 to 15th May 2020.
  register and compare the ICU admission between both periods.
Register the Hospital stay | PreCOVID group from 13th January 2020 to 29th February 2020 and COVID group from 11th March 2020 to 15th May 2020.
  register and compare the ICU admission between both periods.
Register the Mortality | PreCOVID group from 13th January 2020 to 29th February 2020 and COVID group from 11th March 2020 to 15th May 2020.
  register and compare the Mortality between both periods.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jose MJ Colomina, PhD, Principal Investigator — Head of the Department
Locations (1):
- Marta Caballero, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Caballero-Milan M, Colomina MJ, Marin-Carcey LA, Viguera-Fernandez L, Bayona-Domenge R, Garcia-Ballester S, Lopez-Farre A, Ruiz-Buera L, Sanz-Iturbe M, Alvarez-Villegas D, Jenssen-Paz EC, Puig-Sanz G, Arcos-Terrones A, Belmonte-Cuenca C, Perelada-Alonso E, Blasco-Blasco F, Sabate A. Impact of the SARS-CoV-2 (COVID19) pandemic on the morbidity and mortality of high risk patients undergoing surgery: a non-inferiority retrospective observational study. BMC Anesthesiol. 2021 Nov 26;21(1):295. doi: 10.1186/s12871-021-01495-3. PMID 34836504

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/94/NCT04780594/Prot_SAP_000.pdf